CLINICAL TRIAL: NCT05706506
Title: An Open-Label, Single-Arm, Phase 4 Study to Assess Glycemic Control When Adults With Type 2 Diabetes Switch From a GLP-1 RA to Tirzepatide (SURPASS-SWITCH-2)
Brief Title: A Study of Tirzepatide (LY3298176) in Adults With Type 2 Diabetes Switching From a GLP-1 RA (SURPASS-SWITCH-2)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18520; I8F-MC-GPIL (Other: Eli Lilly and Company); 2022-002708-18 (EudraCT Number)
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 5 milligrams (mg) Tirzepatide (Experimental): Participants received 5 mg tirzepatide subcutaneously administered once weekly for 12 weeks.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176

SUMMARY:
The main purpose of this study is to investigate the effects of switching from glucagon-like peptide-1 receptor agonist (GLP-1 RA) therapy to tirzepatide glucose-dependent insulinotropic polypeptide (GIP) GLP-1 RA agonist in participants with type 2 diabetes (T2D).

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 diabetes (T2D)
* Have an HbA1c c ≥6.5% (≥48 mmol/mol) to ≤9.0% (≤75 mmol/mol)
* Have a body mass index (BMI) ≥25 kilogram per square meter (kg/m²) at screening
* Have been on a stable treatment dose of 1 of the listed GLP-1 RAs for ≥3 months
* No treatment with oral antidiabetic medicine (OAM) or on stable doses (for at least 3 months before screening) of up to 3 OAM. The OAM may include metformin, sodium-glucose linked transporter-2 inhibitor (SGLT-2i), thiazolidinediones, or α-glucosidase inhibitors.

Exclusion Criteria:

* Have Type 1 Diabetes (T1D)
* Have a clinical history of

  * proliferative diabetic retinopathy
  * diabetic maculopathy, or
  * non-proliferative diabetic retinopathy that requires acute treatment
* Are at high risk for cardiovascular disease or have a history of

  * myocardial infarction
  * percutaneous coronary revascularization procedure
  * carotid stenting or surgical revascularization
  * nontraumatic amputation
  * peripheral vascular procedure
  * cerebrovascular accident
  * or hospitalization for congestive heart failure
* Have New York Heart Association (NYHA) Functional Classification Class IV congestive heart failure
* Have a history of ketoacidosis or hyperosmolar state or coma
* Have a history of severe hypoglycemia or hypoglycemia unawareness within the 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (32):
- United States (32):
  - Fiel Family and Sports Medicine PC, Tempe, Arizona
  - New Hope Research Development, Corona, California
  - Velocity Clinical Research, Gardena, Gardena, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Velocity Clinical Research, Huntington Park, Los Angeles, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Dream Team Clinical Research, Pomona, California
  - Scripps Whittier Diabetes Institute, San Diego, California
  - Metabolic Institute of America, Tarzana, California
  - CMR of Greater New Haven, LLC, Waterbury, Connecticut
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Florida Institute For Clinical Research, LLC, Orlando, Florida
  - New Tampa Health, Tampa, Florida
  - Georgia Clinical Research, Lawrenceville, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Velocity Clinical Research, Valparaiso, Valparaiso, Indiana
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Clinic, Topeka, Kansas
  - Versailles Family Medicine, Versailles, Kentucky
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - Clinical Research Professionals, Chesterfield, Missouri
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - Advanced Medical Research, Maumee, Ohio
  - Conrad Clinical Research, Edmond, Oklahoma
  - Mountain View Clinical Research, Inc., Greenville, South Carolina
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Memorial City Endocrine Consultants, Houston, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - ClinPoint Trials, Waxahachie, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org

REFERENCES:
- See also: A Study of Tirzepatide (LY3298176) in Adults With Type 2 Diabetes Switching From a GLP-1 RA (SURPASS-SWITCH-2) — https://trials.lilly.com/en-US/trial/385077

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 Milligrams (mg) Tirzepatide: Participants received 5 mg tirzepatide subcutaneously (SC) administered once weekly (QW) for 12 weeks.
Period: Overall Study
Arm/Group | 5 Milligrams (mg) Tirzepatide
Started | 152
Received At Least 1 Dose of Study Drug | 152
Completed | 131
Not Completed | 21
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 2
Not completed — Inadvertent Enrolment | 12
Not completed — Early Discontinuation Due to Hyperglycemia | 1
Not completed — Participant Moved Out of State | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of tirzepatide.
Groups:
- 5 mg Tirzepatide: Participants received 5 mg tirzepatide SC administered QW for 12 weeks.
Arm/Group | 5 mg Tirzepatide
Number analyzed (Participants) | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32
  Not Hispanic or Latino | 120
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 117
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 152
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 7.40 (0.660)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Baseline, Week 12
Population: All participants who received at least one dose of tirzepatide, had a baseline and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 5 mg Tirzepatide
Number analyzed (Participants) | 140
Percentage of HbA1c | -0.43 (0.05)

2. Secondary Outcome: Change From Baseline in Percentage of Time Per Day That Continuous Glucose Monitoring (CGM)-Derived Values Were >180 Milligram/Deciliter (mg/dl) (10 Millimole/Liter (mmol/L))
Description: Change from Baseline in Percentage of Time per Day that CGM-derived Values were >180 mg/dl (10 mmol/L) was assessed.
Time Frame: Baseline, Week 4
Population: All participants who received at least one dose of tirzepatide, had a baseline and at least one post-baseline value for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Percentage of time per day
Arm/Group | 5 mg Tirzepatide
Number analyzed (Participants) | 140
Percentage of time per day | -6.52 (1.55)

3. Secondary Outcome: Change From Baseline in Percentage of Time Per Day That CGM-derived Values Were >180 mg/dl (10 mmol/L)
Description: Change from Baseline in Percentage of Time per Day that CGM-derived Values were >180 mg/dl (10 mmol/L) was assessed.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of time per day
Arm/Group | 5 mg Tirzepatide
Number analyzed (Participants) | 140
Percentage of time per day | -7.37 (1.54)

4. Secondary Outcome: Change From Baseline in Duration of Time in Minutes Per Day That CGM Derived Values Were >180 mg/dl (10 mmol/L)
Description: Change from Baseline in Duration of Time in Minutes per Day that CGM derived Values were >180 mg/dl (10 mmol/L) was assessed.
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Minutes per day
Arm/Group | 5 mg Tirzepatide
Number analyzed (Participants) | 140
Minutes per day | -93.82 (22.30)

5. Secondary Outcome: Change From Baseline in Duration of Time in Minutes Per Day That CGM Derived Values Were >180 mg/dl (10 mmol/L)
Description: as for outcome 4
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Minutes per day
Arm/Group | 5 mg Tirzepatide
Number analyzed (Participants) | 140
Minutes per day | -106.09 (22.21)

6. Secondary Outcome: Change From Baseline in Fasting Serum Glucose (FSG)
Description: Change from Baseline in FSG was assessed.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | 5 mg Tirzepatide
Number analyzed (Participants) | 140
milligrams per deciliter (mg/dL) | -7.83 (2.85)

7. Secondary Outcome: Change From Baseline in Weight
Description: Change from Baseline in Weight was assessed.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 5 mg Tirzepatide
Number analyzed (Participants) | 140
kilograms (kg) | -2.15 (0.28)

ADVERSE EVENTS:
Time Frame: Baseline Up To 12 Weeks
Description: All participants who received at least one dose of tirzepatide.
Arm/Group | 5 mg Tirzepatide
All-Cause Mortality (participants affected / at risk) | 0/152
Serious Adverse Events (participants affected / at risk) | 1/152
Other Adverse Events (participants affected / at risk) | 0/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tirzepatide (N=152)
Coronary artery disease (Cardiac disorders) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT05706506/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT05706506/SAP_001.pdf